CLINICAL TRIAL: NCT03300154
Title: Effectiveness of Financial Incentives and Text Messages to Improve Health Care of Vulnerable Population With Moderate and High Cardiovascular Risk in Argentina: A Randomized Cluster Trial
Brief Title: Effectiveness of Financial Incentives and Text Messages to Improve Health Care in Population With Moderate and High Cardiovascular Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AR-T1087-P0001/2
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Moderate and High Cardiovascular Risk
Keywords: Cardiovascular risk; Behavioral economics; Text messages; Financial incentives
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Financial incentives (Experimental)
  Interventions: Behavioral: Financial incentives
- Framing (SMS) (Experimental)
  Interventions: Behavioral: Framing (SMS)
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Financial incentives — The study nurses will schedule an appointment with the doctor at the health center, within 4 weeks from the participant's inclusion in the study. Participants who attend the first visit at the health center will receive a direct incentive consisting of the payment of a limited amount to be determined (approximately AR $ 150-200) through a shopping voucher for the amount mentioned. Participants attending the follow-up visit at the health center within 3 months from their inclusion in the study will participate in a lottery. The lottery will offer the possibility of winning a new voucher with a probability of 1 in 3. Participants who do not attend the health center will not receive any incentive.
  Arms: Financial incentives
Behavioral: Framing (SMS) — After inclusion, participants will receive weekly text messages (SMS) using a specific framing or formulation of the message, highlighting the potential benefits and positive aspects of health care. These messages will promote follow-up visits, adherence to treatment, and benefits to be gained from a follow-up visit with the physician. Messages will be sent with a frequency of two per week during the first 30 days and then 1 per week until the end of the follow-up. These messages will have no cost to participants.
  Arms: Framing (SMS)

SUMMARY:
Cardiovascular diseases are increasing throughout the developing world and are the cause of almost 16.7 million deaths each year, of which 80% occur in low and middle-income countries. As more than three fourth of the global burden of cardiometabolic diseases are related to risk factors connected with lifestyles or behaviors, such as smoking, unhealthy eating, low physical activity, and harmful consumption of alcohol. This burden could be dramatically reduced by changing individual behaviors. This study is focused on interventions that are aimed to improve the adherence to treatment in cardiovascular disease (hypertension), based on a Behavioral Economics approach. Most of public policies targeted to tackle NCDs utilize a rational economic model of behavior. Behavioral economics, by using insights from cognitive psychology and other social sciences, has drawn a lot of attention for its potential to increase healthy behaviors. Interventions informed by BE principles seek to rearrange the social or physical environment in such a way to 'nudge' people towards healthier choices and behaviors.

Main objective: to assess whether the implementation of two strategies based on behavioral economics, that include the use of a financial incentive scheme and specific framing to beneficiaries (i.e. mobile health interventions), increase the referral, evaluation and follow-up of people with moderate and high cardiovascular risk in the public health network, compared to the usual strategy.

Design: A cluster-randomized pragmatic clinical trial will be performed. The randomization unit will be the Community Health Centers (CHC) and the intervention groups (2 arms) or control will be assigned to 9 health centers in total (3 CHC per arm).

Population: This RCT is going to be conducted in selected CHC of Salta. Nine CHC will be selected, which will be randomized: 3 centers to the control, 3 centers to framing intervention with messages and 3 centers to the intervention with incentives.

A total of 900 patients ≥ 40 years, without health coverage and with a 10-year cardiovascular risk ≥ 10% will participate in this study.

Follow up: 3 month

ELIGIBILITY:
Inclusion Criteria:

* Subjects that only have public health coverage.
* Residence in the area of influence of the health centers of the study.
* Have a mobile phone for personal use.
* 10 year cardiovascular risk ≥ 10%

Exclusion Criteria:

* Pregnant women.
* Immobilized people.
* Persons who do not give their informed consent.
* People planning to move in the next 3 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 917 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-10-23 (Estimated)

PRIMARY OUTCOMES:
Attendance at the first medical visit | 4 weeks
  Proportion of patients who attended and completed the first clinical visit to the health center
Attendance at the second medical visit | 8 weeks after first medical visit
  Proportion of patients who attended and completed the second clinical visit to the health center

SECONDARY OUTCOMES:
Attendance at least one clinical visit | 12 weeks
  Proportion of patients who attended and completed at least one clinical visit to the health

CONTACTS AND LOCATIONS:
Locations (9):
- Argentina (9):
  - 1º DE MAYO, General Güemes, Salta Province
  - Barrio Cooperativa, General Güemes, Salta Province
  - Barrio La Tablada, General Güemes, Salta Province
  - Campo Santo, General Güemes, Salta Province
  - CIC, General Güemes, Salta Province
  - EL BORDO, General Güemes, Salta Province
  - El cruce, General Güemes, Salta Province
  - Los Olivos, General Güemes, Salta Province
  - Villa Tranquila, General Güemes, Salta Province

REFERENCES:
- [Derived] Poggio R, Prado C, Santero M, Nejamis A, Gutierrez L, Irazola V. Effectiveness of financial incentives and message framing to improve clinic visits of people with moderate-high cardiovascular risk in a vulnerable population in Argentina: A cluster randomized trial. Prev Med. 2021 Dec;153:106738. doi: 10.1016/j.ypmed.2021.106738. Epub 2021 Jul 20. PMID 34298028